Follow the sutures. A new procedure for injection of Botulinum Toxin for Chronic Migraine.

Statistical Analysis Plan

Version 1.0

# 1. Administrative information

| Sponsor name | St. Olavs Hospital |
|---|---|
| Sponsor address | Nevroklinikken, 7006 Trondheim, Norway |
| Unique protocol ID (Ethics approval) | 2017/1490 |
| Secondary IDs (EUDRACT) | 2017/002516-13 |
| ClinicalTrials.gov | NCT03543254 |
| Trial title | Follow the sutures. A new procedure for |
| | injection of Botulinum Toxin for Chronic |
| | Migraine. |

SAP and protocol version

| SAP version and date | This SAP is version 1, dated January 8, 2024 |
|----------------------|----------------------------------------------|
| Protocol version | This document was written based on |
| | information contained in the study protocol |
| d d | version 1.0, March 20, 2018 |

SAP revision history

| Protocol version | SAP version | Section number changed | Description and reason for | Date changed |
|---|---|---|---|---|
| | | South | change | |
| | 1.0 | | First edition of | |
| | | | SAP | fs. |

# 2. Signature page

Principal investigator:

Knut Hagen, MD, PhD

Department of Neurology, St. Olavs University Hospital, 7006 Trondheim, Norway Norwegian University of Science and Technology (NTNU) Trondheim, Norway

Signature

Date (08/01/2024)

## 3. Abbreviations

| PREEMT studies | ClinicalTrials.gov |
|----------------|-----------------------------------------------------|
| | identifiers <u>NCT00156910</u> , <u>NCT00168428</u> |

# Table of contents

| Title | | ert. |
|-------|----------------------------------------------------------|-----------|
| 2. S | gnature page | 2 |
| 3. A | bbreviations | 3 |
| 4. Iı | troduction | 6 |
| 4 | 1 Background and rationale | 6 |
| 4 | 2 Trial objectives | 6 |
| | 4.2.1 Primary objective | 6 |
| | 4.2.2 Secondary objectives | |
| 4 | 3 Trial endpoints | |
| | 4.3.1 Primary endpoints | |
| | • | |
| | r <b>ial methods</b> | |
| | 1 Trial design | |
| 5 | 2 Randomization | 6 |
| 5 | 3 Sample size | 6 |
| 5 | 4 Statistical framework | 6 |
| | 5.4.1 Hypothesis test | 6 |
| | 5.4.2 Statistical interim analyses | |
| | 5.4.3 Timing of final analysis | |
| | 5.4.4 Endpoint assesments | /<br>ert. |
| 5 | 5 Blinding procedure | |
| | atistical principles | |
| 6 | 1 Confidence intervals and p-values | 7 |
| 6 | 2 Adherence, protocol deviations and protocol violations | 7 |
| | 6.2.1 Headache diary adherence | 7 |
| | 6.2.2.Protocol violations | |
| 6 | 3 Analysis populations | 7 |
| 7. T | rial population | 7 |
| | 1 Screening data, eligibility, and recruitment | |
| | 2 Withdrawal/Lost to follow-up | |
| / | 3 Baseline patient characteristics | / |
| 8. A | nalysis | 7 |
| 8 | 1 Analysis of the primary efficacy endpoint | 8 |
| | 8.1.1 Statistical methods | |
| | 8.1.2 Missing data | 8 |
| 8 | 2 Analysis of the secondary endpoints | 8 |
| | 8.2.1 Missing data | 8 |
| 8 | 3 Subgroup analyses | 8 |
| 0 5 | foty Analyses | Q |

| 10 | Statistical Software | Q |
|----|------------------------------------|---|
| | 9.3 Vital Signs | 8 |
| | 9.2 Clinical Laboratory Parameters | 8 |
| | 9.1 Adverse Events | 8 |

#### 4. Introduction

### 4.1 Background and rationale

The preclinical data suggest that a "follow-the-suture" approach to injections of onabotulinumtotoxin-A in patients with chronic migraine could represent an effective and less invasive and costly injection strategy than the currently employed pooled analysis of two large studies (PREEMPT-1 and 2) injection paradigm. The aim of the present pilot study was to develop a follow-the-suture injection paradigm and evaluate its feasibility, tolerability, and acceptability among patients with chronic migraine in an open-label pilot study

### 4.2 Trial objectives

### 4.2.1 Primary objective

The primary objective was to develop a follow-the-suture injection paradigm

### 4.2.2 Secondary objectives

Secondary objectives were to evaluate feasibility, tolerability, and acceptability among patients with chronic migraine in an open-label pilot study

### 4.3 Trial endpoints

### 4.3.1 Primary endpoints

• The primary endpoint was number of adverse events recorded during the study.

### 4.3.2 Secondary endpoints

- Compared to baseline, change in weeks 5–8 of: moderate/severe headache days (main efficacy variable), defined as headache lasting >4 h with at least moderate intense pain;
- Compared to baseline, change in weeks 5–8 of headache days, defined as a day with headache lasting >4 h with mild, moderate, or severe pain;

### 5.1 Trial design

An open-label pilot study

#### 5.2 Randomization

No randomization was performed.

#### 5.3 Sample size

Twenty patients with chronic migraine were included, all women.

#### 5.4 Statistical framework

#### 5.4.1 Hypothesis test

The null hypothesis is that there is no difference in of adverse events compared to previous employed pooled analysis of two large studies (PREEMT 1 and 2).

#### 5.4.2 Statistical interim analyses

No interim analysis was performed in this pilot study.

### 5.4.3 Timing of final analysis

Adverse events was collected during the 3-month follow-up. Headache at baseline was compared to weeks 5–8 of follow-up.

### 5.4.4 Endpoint assessments

### 5.4.4.1 Headache diary

Patients were then given instructions in completion of a paper headache diary, where they recorded pain intensity and duration, concomitant migraine symptoms (nausea, vomiting, phono- and photophobia), acute medication (type, number of doses) and work absence (yes/no/not relevant). In addition, they were asked to record any adverse events.

### 5.5 Blinding procedure

The study is open-labelled.

### 6. Statistical principles

### 6.1 Confidence intervals and p-values

Statistically significant change from baseline was tested with a paired t-test. P < 0.05 was considered significant.

### 6.2 Adherence, protocol deviations and protocol violations

### 6.2.1 Headache diary adherence

The participant will be separated into two groups, filled in a headache diary and not filled in a headache diary

#### 6.2.2. Protocol violations

Only number with complete data will be presented for each variable. No participant had protocol violation.

### 6.3 Analysis populations

The 20 participants with written consent

## 7. Trial population

### 7.1 Screening data, eligibility, and recruitment

Only patients with signed written consent will be reported.

### 7.2 Withdrawal/Lost to follow-up

Non patients with withdrawal or lost to follow-up

### 7.3 Baseline patient characteristics

The gender distribution, mean age, and use of acute and preventive medication will be given.

#### 8. Analysis

### 8.1 Analysis of the primary efficacy endpoint

The primary outcome is number of adverse events recorded during the study. This will be given in a Table divided by timing of follow-up (baseline period, week 1-4, week 5-8, and week 9-12.

#### 8.1.1 Statistical methods

Number of participants with adverse events will be given in each study period without statistical comparison.

### 8.1.2 Missing data

No data will be discarded.

### 8.2 Analysis of the secondary endpoints

For the secondary efficacy variables, mean values with standard deviations for each 4-week period, change (in %) between baseline and each 4-week period, and the whole 12-week period after injection were calculated. In patients who had recorded more than 4 weeks in the baseline period, only the first 28 days were considered. In the protocol, the secondary efficacy endpoint was defined as the change in week 5–8

### 8.2.1 Missing data

Missing data for secondary outcomes will not be imputed in this study.

### 8.3 Subgroup analyses

No subgroup analyses will be performed

### 9. Safety Analyses

#### 9.1 Adverse Events

All adverse events and other health issues are registered in the paper version of the headache diary.

### 9.2 Clinical Laboratory Parameters

Not applicable.

### 9.3 Vital Signs

Not applicable.

#### 10. Statistical Software

All statistical analyses will be done using SPSS version 27 (IBM corp., Chicago, IL).